CLINICAL TRIAL: NCT02210962
Title: Omega-3 Fatty Acids in First-episode Schizophrenia - a Randomized Controlled Study of Efficacy and Relapse Prevention (OFFER). Rationale, Design, and Methods.
Brief Title: Omega-3 Fatty Acids Efficacy in First-episode of Schizophrenia
Acronym: OFFER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Tomasz Pawelczyk, Assistant Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N N402 243435
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: early psychosis; chronic schizophrenia; first episode psychosis; omega-3 and omega-6 essential fatty acids; relapse prevention; efficacy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Fatty Acids, Essential; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- essential fatty acids (Experimental): The experimental treatment is a food supplement containing fish oil. The daily dose of 4 capsules provides 1320 mg of eicosapentaenoic acid and 880 mg of docosahexaenoic acid, 26 weeks intervention
  Interventions: Dietary Supplement: essential fatty acids
- olive oil (Placebo Comparator): Placebo capsules contain olive oil and trace amount of fish oil to assure comparable taste, 26 weeks intervention
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: essential fatty acids — Yellow capsules containing eicosapentaenoic acid, docosahexaenoic acid (active)
  Arms: essential fatty acids
Dietary Supplement: olive oil — Yellow capsules containing olive oil (placebo)
  Arms: olive oil

SUMMARY:
There is accumulating experimental evidence to suggest the role of essential fatty acids (EFA) in neuronal migration, pruning and synaptic plasticity. These processes are implied to be dysfunctional on early stages of schizophrenia, according to neurodevelopmental hypothesis. Numerous epidemiological and clinical trial data support the benefit of EFA rich diets in reducing symptoms in schizophrenia. An EFA rich diet might be of particular importance at the beginning of the illness. As a relatively safe option, EFA supplementation would be a preferable add on therapy in treating individuals with a first episode of schizophrenia (FES) and a short duration of psychotic symptoms. No long term follow-up studies of EFA supplementation in FES patients were carried out. The demonstration of the efficacy of the prophylactic properties of EFAs in relapse prevention in FES patients would be a strong basis for further studies and prescribing EFAs for a large population of patients who are in the early stages of that debilitating illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia using Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria
* Patients aged between 16-35 years
* Signed informed consent (parallel parents consent for individuals under 18 years of age)

Exclusion Criteria:

* Patients taking fish oil supplements (a washout period of 6 months is required)
* Patients diagnosed with epilepsy or suffering from epileptic seizures
* Patients receiving anticoagulant medication e.g., Warfarin
* Patients receiving psychotherapy
* Chronic somatic diseases
* Psychoactive substance dependence
* Pregnancy and lactation
* Mental retardation or diagnosed organic brain injury

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the efficacy of n-3 PUFA in reducing psychopathology in first-episode schizophrenia. | 8 and 26 weeks of supplementation
  The Positive and Negative Syndrome Scale [64] will be used to assess the efficacy of EPA+DHA supplementation in reducing symptom severity in first-episode schizophrenia after 8 and 26 weeks of supplementation. The main outcome measure will be the change in symptom severity from baseline to week 26. Baseline PANSS total score will be subtracted from PANSS score obtained after 26 weeks, resulting in the degree of change observed in the study.

SECONDARY OUTCOMES:
Relapse rate - Positive and Negative Syndrome Scale (PANSS) defined schizophrenia relapse | 26 weeks intervention plus 26 weeks observation
PANSS total, positive, negative and general psychopathology subscales | Baseline, 1, 2, 4, 6, 8, 16, 26, 52 weeks
Calgary Depression Scale for Schizophrenia (CDSS) | Baseline, 1, 2, 4, 6, 8, 16, 26, 52 weeks
Clinical Global Impression (CGI) | Baseline, 1, 2, 4, 6, 8, 16, 26, 52 weeks
Global Assessment of Functioning (GAF) | Baseline, 1, 2, 4, 6, 8, 16, 26, 52 weeks
A white matter directional organization metric: fractional anisotropy (FA) measured in two areas: corpus callosum and uncinate fasciculus | Baseline, 26 weeks
Cognitive performance using composite battery of neuropsychologic tests | Baseline, 8 and 26 weeks
Niacin Flush Skin Test | Baseline, 8 and 26 weeks
Side effects profile according to self-prepared questionnaire | Baseline, 4, 8, 26
Lymphocyte telomerase activity | Baseline, 8 and 26 weeks
Equivalent doses of antipsychotics used | Baseline, 1, 2, 4, 6, 8, 16, 26 and 52 weeks
Grey matter volume: a voxel based structural MRI assessment | Baseline, 8 and 26 weeks

OTHER OUTCOMES:
Plasma cholesterol and Triglycerides | Baseline, 1, 2, 4, 6, 8, 26 and 52 weeks
Blood pressure | Baseline, 1, 2, 4, 6, 8, 26 and 52 weeks
Body mass index (BMI) | Baseline, 1, 2, 4, 6, 8, 26 and 52 weeks
Waist circumference | Baseline, 1, 2, 4, 6, 8, 26 and 52 weeks
Fasting glucose levels | Baseline, 1, 2, 4, 6, 8, 16, 26, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz P Pawełczyk, MD, PhD, Principal Investigator — Department of Affective and Psychotic Disorders Medical University of Lodz
Locations (1):
- Department of Affective and Psychotic Disorders Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

REFERENCES:
- [Derived] Pawelczyk T, Grancow M, Kotlicka-Antczak M, Trafalska E, Gebski P, Szemraj J, Zurner N, Pawelczyk A. Omega-3 fatty acids in first-episode schizophrenia - a randomized controlled study of efficacy and relapse prevention (OFFER): rationale, design, and methods. BMC Psychiatry. 2015 May 2;15:97. doi: 10.1186/s12888-015-0473-2. PMID 25934131